CLINICAL TRIAL: NCT03052413
Title: Study to Evaluate Safety and Efficacy of a Nutraceutical Supplement With Standardized Botanicals for Treatment of Hair Loss and Thinning in Females
Brief Title: Study to Evaluate a Nutraceutical Supplement for Treatment of Hair Loss and Thinning in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sadick Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRG-Nutra-01
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Hair Loss
Keywords: thinning hair; female pattern hair loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Dietary Supplement: Nutrafol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Nutrafol — Eligible subjects will receive Nutrafol® to take daily for 180 days
  Arms: Active
Dietary Supplement: placebo — Eligible subjects will receive Placebo to take daily for 180 days
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the safety and effectiveness of a nutraceutical supplement for the treatment of hair loss and thinning in females over the course of six months of continuous daily use.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, study in adult female subjects with mild to moderate hair loss. Following an up to 35-day screening period to determine eligibility, subjects will be randomly assigned into one of the following treatment arms: Nutrafol® vs. Placebo. Nutrafol® or Placebo will randomly assigned be administered daily to the subjects for 6 months starting on Day 2. The subjects will return to the study site at Day 90 and Day 180 for assessments. Additionally, the subjects will return to the study site approximately 48 hours after Day 0 (Baseline Visit) and D180 in order to assess hair growth rate. Nutrafol® or Placebo will be dispensed by the non-blinded study staff with nonlabeled containers containing the corresponding tablets. Efficacy ratings will be performed by a trained investigator who will not be aware of the subject's treatment randomization in order to preserve double-blinding of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Females between 21 - 55 years of age, inclusive
2. Skin type I-IV
3. Have self-reported thinning or hair loss for more than 6 months prior to screening
4. Clinically confirmed to have hair loss or thinning by the investigator via physical exam, including subjects with female pattern hair loss with Savin Classification score of I2-II1 as determined by the investigator (through medical history, physical exam and /or strong family history of hair loss as defined by 2 or more relatives known to have a similar Savin pattern of loss without diagnosed disease)
5. In good general health, as determined by the Investigator
6. Willing and able to attend all study visits
7. Willing to maintain the same hair style as at the Screening Visit for the duration of the study. If coloring hair, willing to color it with the same frequency of usage as in the past, making sure not to color within 3 weeks of an in-office appointment.
8. Willing to use a mild non-medicated shampoo and conditioner for the duration of the study (medicated shampoo and conditioner refer to any prescription shampoo or conditioner as well as any over-the counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth)
9. Willing to have their hair clipped and scalp tattoo
10. Have a negative urine pregnancy test at screening and be using, and continue to use for the duration of the study, an effective contraception method (ie, abstinence, barrier control, intrauterine device [IUD], or hormonal [estrogen/progestin] contraceptives) for at least one menstrual cycle prior to study; if using IUD or hormonal contraceptives - then at least 2 years prior to screening, the initiation of which should not have been associated with initiation of hair loss/thinning.
11. Be willing and able to cooperate with the requirements of the study.
12. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board.
13. Be able to complete and understand the various rating instruments in English.
14. Sponsor approved global image assessment of degree of thinning / hair loss

Exclusion Criteria:

1. Clinical diagnosis of alopecia areata or scarring forms of alopecia
2. Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
3. Subjects who are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy, or Subjects of childbearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as postmenopausal (absence of menstrual bleeding for one year), hysterectomy or bilateral oophorectomy.
4. Current skin disease (e.g., psoriasis, atopic dermatitis, skin cancer, eczema, sun damage, seborrheic dermatitis), cuts and or abrasions on the scalp or condition (e.g., sunburn, tattoos) on the treatment area that, in the opinion of the Investigator, might put the subject at risk or interfere with the study conduct or evaluations.
5. History of surgical correction of hair loss on the scalp/ Hair transplants.
6. Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within the 30 days prior to the Baseline Visit.
7. Use of anti-androgenic therapies (e.g., spironolactone, flutamide, cyproterone acetate, cimetidine) within 30 days prior to the Baseline Visit.
8. No history of burning, flaking, itching, and stinging of the scalp.
9. History of malignancy (except scc and bcc skin cancers) or undergoing chemotherapy or radiation treatments.
10. A known history of autoimmune thyroid disease, any other thyroid disorder/abnormality or other autoimmune disorders that in the opinion of the investigator may interfere with the study treatment.
11. A known history of depression or bi-polar disease or any other condition that may impact the subject's participation.
12. Subjects taking vitamin E supplements can participate, provided medication is interrupted 14 days before baseline visit.
13. Recent utilization of low level lasers.
14. Has any condition that the treating investigator or PI thinks may put the Subject at risk or interfere with their participation in the study.
15. Is involved in any injury litigation claims
16. Known history or recent bloodwork indicating iron deficiency, bleeding disorders or platelet dysfunction syndrome as well as subjects receiving anticoagulant therapy or smokers with usage >20 cigarettes/day.
17. Use of any medications that are known to potentially cause hair loss or affect hair growth, as determined by PI.

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
change in hair density | 180 days
  change in hair density over the course of the study assessed by hair count

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Sadick Research Group, New York, New York